CLINICAL TRIAL: NCT00992303
Title: Tissue Procurement and Outcome Collection for Radiotherapy Treated Patients and Healthy Participants
Brief Title: Collecting Tissue Samples From Patients With Cancer Undergoing Radiation Therapy and Healthy Participants
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Timmerman, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 072010-098; SCCC-032009-049; CDR0000653406
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: biologic sample preservation procedure
Other: medical chart review
Other: questionnaire administration

SUMMARY:
RATIONALE: Collecting and storing samples of tissue from patients with cancer to test in the laboratory may help the study of cancer in the future.

PURPOSE: This research study is collecting tissue samples from patients with cancer undergoing radiation therapy. Healthy participants will also be allowed on the trial so their samples can be used in comparison to patients with malignancy

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To maintain and create a University of Texas Southwestern Medical Center (UTSW) Radiation Oncology Tissue Resource and Registry/Database that will be used to explore genetic variations contributing to clinical outcomes through tissue analysis and outcome correlation. Tissue will be stored by the UTSTR and the database managed by Radiation Oncology.

Secondary

* To document disease outcome (local recurrence, distant metastasis, overall survival) by treatment regimen and disease site.
* To document toxicity by treatment regimen and disease site.
* To establish a prospective registry/database consisting of patient demographics and outcomes to be used for future research.

OUTLINE: Tissue, including surgical waste, venous blood/serum, urine, bone marrow, and other body fluids, may be collected (at planned surgery and routine medical visits) and preserved for future research. Demographic and disease and treatment information is obtained from patients (by interview or questionnaire), from medical records, and from national datasets. Patients may also be asked to provide additional blood samples and/or a small skin-punch biopsy sample.

Patients are followed up every 6 months for the first two years following treatment and then yearly thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically-proven diagnosis of malignancy
* Planning treatment with radiation therapy

PATIENT CHARACTERISTICS:

* Able to perform follow-up visits
* Is a patient of the University of Texas Southwestern Medical Center physicians

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Participation in other clinical trials is allowed
* Other prior or concurrent therapy for cancer, such as surgery and/or chemotherapy, is allowed.

Criteria for eligibility:

* Able to provide written informed consent
* Age greater than 18 years old
* Males and Females are eligible
* Any ethnicity is eligible

Criteria for ineligibility:

-Patients not available for follow-up/future contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer patients, healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2009-09; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Maintenance a Tissue Resource and Registry/Database | 10 years
  Maintenance and creation of a University of Texas Southwestern Medical Center (UTSW) Radiation Oncology Tissue Resource and Registry/Database

SECONDARY OUTCOMES:
Local recurrence | 5 years
  To document local recurrence by treatment regimen and disease site.
Distant metastasis | 5 years
  To document distant metastasis by treatment regimen and disease site.
Overall survival | 5 years
  To document overall survival by treatment regimen and disease site.
Toxicity by treatment regimen | 1 year
  To document toxicity by treatment regimen and disease site.
Establishment of a prospective registry/database | 10 years
  To establish a prospective registry/database consisting of patient demographics and outcomes to be used for future research.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Timmerman, MD, Principal Investigator — University of Texas Southwestern Medical Center - Dallas
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States